CLINICAL TRIAL: NCT06971653
Title: Piezoelectric Versus Conventional Surgical Approaches in Third Molar Removal: A Focus on Pain, Comfort, and Patient Satisfaction
Brief Title: Effect of Piezoelectric Surgery on Pain, Comfort, and Patient Satisfaction in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mert Zeytinoğlu, Assoc. Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGE-DHF-MZ-004
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Oral Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 patients in the piezoelectric surgery group (Experimental)
  Interventions: Procedure: piezoelectric surgery
- 30 patients in the conventional surgery group (Experimental)
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: conventional surgery — This retrospective clinical study included 30 patients who underwent extraction of impacted lower third molars with conventional surgery
  Arms: 30 patients in the conventional surgery group
Procedure: piezoelectric surgery — This retrospective clinical study included 30 patients who underwent extraction of impacted lower third molars with piezoelectric surgery
  Arms: 30 patients in the piezoelectric surgery group

SUMMARY:
The purpose of this study is to compare the effects of piezoelectric surgery on postoperative pain, comfort and patient satisfaction with conventional bur method applied in surgical extraction of impacted mandibular third molars.

The main question it aims to answer is:

Is piezoelectric surgery effective on reducing pain and increasing comfort and patient satisfaction in impacted third molar surgery? Pain levels were assessed using the Visual Analog Scale (VAS), and patient satisfaction was measured with functional evaluations conducted on the 1st, 3rd, and 7th postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mesioangular, distoangular, vertical or horizontal, fully impacted and fully bone retained impacted lower wisdom teeth
* Patients without any systemic disease
* Patients who have been informed about the duration, purpose and requirements of the study and who have signed the informed consent form voluntarily.

Exclusion Criteria:

* Patients with any systemic contraindication, infection in the area of the tooth to be extracted, anamnesis of sensitivity to paracetamol derivatives or aspirin, pregnant or breastfeeding patients, and patients using antibiotics or anti-inflammatory drugs in the last 3 weeks
* In addition, smokers or alcohol addicts were not included in the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain with Routine and Piezoelectric Surgery | The postoperative outcomes including pain are clinically assessed at different-time intervals (6th and 12th hours after the operation, 1st, 2nd, 3rd and 7th days after the operation).
  The primary outcome measure is postoperative pain with Routine and Piezoelectric Surgery in bilateral impacted third molar. Postoperative pain is assessed using the numbered and visual pain scale. Patients are asked to mark the pain they felt on the scale days after the operation.

SECONDARY OUTCOMES:
Chewing, Swallowing and Speaking Functions with Routine and Piezoelectric Surgery | The postoperative outcomes including chewing, swallowing and speaking are clinically assessed at different-time intervals (1st, 2nd, 3rd, 4th, 5th, 6th and 7th days postoperative days).
  Starting from the first day of the operation until the 7th day when the stitches are removed, the patients mark their subjective complaints about their quality of life on the forms by giving them scores between 0 and 5, considering their chewing, swallowing and speaking functions. (Patient Evaluation Form) These forms are evaluated and the patients' satisfaction with their quality of life is measured in the post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Zeytinoğlu, Principal Investigator — Ege University

IPD SHARING:
Plan to Share IPD: No